CLINICAL TRIAL: NCT01648777
Title: Cicatricial Analgesia Catheters Outcome on Bronchopulmonary Infection Number With Sternotomy Cardiac Operated
Brief Title: Catheter Outcomes With Sternotomy Cardiac Operated
Acronym: STERNOCAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Baxter Healthcare Corporation (Industry); WYM France (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-3289-10; A110903-48 (Other: AFSSAPS)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2013-11

CONDITIONS: Pneumonia; Cardiac Surgery; Multiperforated Catheter; Analgesia; Critical Care Medicine
Keywords: Pneumonia; Postoperative infection; Cardiac surgery; Multiperforated catheter; Analgesia
MeSH Terms: conditions — Pneumonia; Agnosia | interventions — Catheters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L bupivacaine (Experimental): Drug (L bupivacaine) and device (catheter) 750 patients undergoing cardiac surgery with sternotomy are treated with L-bupivacain in the multiperforated catheter of analgesia
  Interventions: Device: L bupivacaine
- placebo (Placebo Comparator): Isotonic Nacl 9°/00 solution 750 patients undergoing cardiac surgery with sternotomy are treated with isotonic NaCl solution (placebo) in the multiperforated catheter of analgesia
  Interventions: Drug: placebo

INTERVENTIONS:
Device: L bupivacaine — L-bupivacain solution CHIROCAINE® 5mg/ml, flakon de 20 ml): for the intravenous bolus of 10 ml
  o (CHIROCAINE®1.25mg/ml, 200 mL/unit, 400 ml in the accufusor infused at 8ml/h during 48h00: for infusion during 48h00
  Other Names: catheter with L bupivacaine
  Arms: L bupivacaine
Drug: placebo — * Isotonic NaCl solution (9°/00) solution: for the intravenous bolus of 10 ml
  * Isotonic NaCl solution (9°/00) solution, 400 ml in the accufusor infused at 8ml/h during 48h00: for infusion during 48h00
  Other Names: Isotonic NaCl solution
  Arms: placebo

SUMMARY:
Pneumonia occurs frequently in patients undergoing cardiac surgery and allows to increase their mortality. While chest physical therapy plays a crucial role to prevent postoperative pneumoniae, painful mobilization of the sternum after sternotomy limits chest physical therapy. The continuous local anesthetic infusion by multiperforated catheter decreases sternum pain. Because of this optimal pain management, early chest physical therapy could be more efficient and could contribute to decrease the rate of pneumonia.

The aim of this study is to test if management of sternotomy pain using continuous local anesthetic infusion by multiperforated catheter may contribute to decrease the rate of perioperative pneumonia.

DETAILED DESCRIPTION:
Introduction:

Pneumonia occurs in 15 to 20% of patients undergoing cardiac surgery and allows to increase their mortality. Early non-invasive ventilation (NIV) after extubation and active and passive chest physical therapies have shown to diminish risk of respiratory failure and lowered 90-day mortality. Unfortunately, pain after cardiac surgery is mainly related to the median sternotomy. The mobilization of the sternum after sternotomy induces paroxysmal and periodical pain, sorely control by opioid treatment, regulated by the chest movements of ventilation or chest mobilization such during NIV or chest physical therapy. The continuous local anesthetic infusion by multiperforated catheter has been shown to be effective for decreasing paroxysmal sternum pain, opioid analgesic medication, length of intensive care medicine (ICU) and hospital stay. Because of this better pain management, early NIV and chest physical therapy could be more efficient and could contribute to decrease the rate of pneumonia in patients undergoing cardiac surgery with sternotomy.

Hypothesis: The aim of this study is to test if management of sternotomy pain using continuous local anesthetic infusion by multiperforated catheter may contribute to decrease the rate of perioperative pneumonia.

Primary end-point: Rate of post-operative pneumonia in hospital. Secondary end-points: post operative quality of Analgesia (total morphine consumption), 30-days all-cause mortality, mechanical ventilation free days, ICU free days, hospital stay, rate of ICU readmission, reintubation rate, septic shock rate, extrarenal epuration rate, cerebral vascular injury rate, Major Cardiac Adverse Events at 30-days, mortality at 30 days.

Method: This is a multicenter (5 french university centers) double blind randomized study compared to placebo. Patients are randomized the day before surgery (computer randomization) between L-bupivacaine and placebo which is infused with continuous local anesthetic infusion by multiperforated catheter at the end of cardiac surgery with sternotomy. Anesthesia protocol is pre-established (propofol and sufentanil with TCI and atracurium only at the induction), tranexamic acid (bolus of 20 mg/kg and 2mg/kg/h). Total dose of each agent is reported in the electronic case report (eCRF, cleanWeb®). Antibioprophylaxy is standardized in agreement with French guidelines in cardiac surgery. Analgesic treatment is standardized as well. During the first postoperative 48 hours: paracetamol (1g x4/day), morphine sulfate (intravenous titration and immediately after the end of titration, self pain management with morphine pump during 48 hours for all the patients included in the study. Total dose of morphine sulfate is reported in the eCRF. In addition, intravenous ketoprofen may be associated in addition if requested. Multiperforated catheter is introduced at the end of surgery above steel sternal bands. A bolus of 10 ml of L-bupivacain or placebo is infused into the catheter at the end of surgery when skin suture is done. Then, the elastomeric pump is connected to the catheter for 48 postoperative hours at 8ml/hour. Extubation is done ideally in the first 6 postoperative hours and chest kinesitherapy is performed at day 1 and 2, in postoperative period. Follow up is done during 30 days after surgery.

Statistical analysis: Rate of pneumonia is expected to be 18% in the placebo group, and 12.6% in the L-bupivacaine group. The number of patients needed (with alpha=0.05, beta= 0.80) is estimated to be 1500 patients (750 patients by group). Because 5 centers are expected to participate, 15% only of eligible patients in all these centers will be enough. Twenty four months would be necessary for the inclusion with 1 month more for the follow up. Thus, the study would last 25 months.

Ethical issue: The present study will be presented to pitie salpetriere Research Ethics Board for approval. An independent Safety Board will survey the study.

Conclusion: This study should decrease the rate of pneumonia in patients undergoing cardiac surgery with sternotomy.

ELIGIBILITY:
Inclusion criteria :

* all patient more than 18 years old
* planned cardiac surgery with sternotomy and bypass
* Informed consent written

Exclusion criteria :

* Refusal of patient to be included in the study
* Age less than 18 years old
* Pregnancy
* Emergency
* Prolonged sedation and ventilation more than 48h00 expected in teh postoperative period
* Moribund patient
* Palliative medicine
* Patient in the care of a guardian
* Preoperative pneumonia
* Patient randomized in an other randomized study
* Contraindication to L-bupivacain, morphine sulfate, paracetamol or tramadol
* Lack of national health care insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1502 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative pneumonia in hospital | 30 days

SECONDARY OUTCOMES:
all-cause mortality | 30 days
mechanical ventilation free days | 30 days
ICU free days | 30 days
Hospital stay | 30 days
Rate of ICU readmission | 30 days
Reintubation rate | 30 days
Septic shock rate | 30 days
Extrarenal epuration rate | 30 days
Cerebral vascular injury rate | 30 days
Major Cardiac Adverse Events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Julien Amour, MD, PhD, Principal Investigator — APHP
Locations (1):
- Pitié salpetrière Hospital, Paris, France

REFERENCES:
- [Derived] Amour J, Cholley B, Ouattara A, Longrois D, Leprince P, Fellahi JL, Riou B, Hariri S, Latremouille C, Remy A, Provenchere S, Carillion A, Achouh P, Labrousse L, Tran Dinh A, Ait Hamou N, Charfeddine A, Lafourcade A, Hajage D, Bougle A; STERNOCAT investigators. The effect of local anesthetic continuous wound infusion for the prevention of postoperative pneumonia after on-pump cardiac surgery with sternotomy: the STERNOCAT randomized clinical trial. Intensive Care Med. 2019 Jan;45(1):33-43. doi: 10.1007/s00134-018-5497-x. Epub 2019 Jan 7. PMID 30617461